CLINICAL TRIAL: NCT01220219
Title: An Open-Label, Multiple-Dose, Randomized, 3-Way Crossover Study In Healthy Volunteers To Determine The Steady-State Pharmacokinetics Of The 82.5 Mg And 165 Mg Dose Strengths Of Pregabalin Controlled Release Formulations Administered Following An Evening Meal And 75 Mg Of The Immediate Release Formulation Administered Twice Daily
Brief Title: An Investigation Of The Absorption And Pharmacokinetics Of Multiple Doses Of Two Controlled Release Pregabalin Tablets As Compared To Multiple Doses Of The Immediate Release Pregabalin Capsule In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081226
Record Dates: First submitted 2010-10-04; First posted 2010-10-13 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2011-01

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability; bioequivalence
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pregabalin controlled release, 82.5 mg (Experimental)
  Interventions: Drug: Pregabalin controlled release, 82.5 mg
- Pregabalin controlled release, 165 mg (Experimental)
  Interventions: Drug: Pregabalin controlled release, 165 mg
- Pregabalin immediate release, 75mg (Other): Reference Treatment
  Interventions: Drug: Pregabalin immediate release, 75mg

INTERVENTIONS:
Drug: Pregabalin controlled release, 82.5 mg — Two tablets of 82.5 mg controlled release (administered concurrently) once daily for four days.
  Arms: Pregabalin controlled release, 82.5 mg
Drug: Pregabalin controlled release, 165 mg — 165 mg controlled release tablet administered once daily for four days.
  Arms: Pregabalin controlled release, 165 mg
Drug: Pregabalin immediate release, 75mg — 75 mg immediate release capsule administered every 12 hours for four days
  Arms: Pregabalin immediate release, 75mg

SUMMARY:
The purpose of this study is to 1) evaluate the extent of absorption of multiple doses of two pregabalin controlled release tablets as compared to multiple doses of the pregabalin immediate release capsule, 2) evaluate the pharmacokinetics of multiple doses of two pregabalin controlled release tablets as compared to multiple doses of pregabalin immediate release capsule and 3) evaluate the safety and tolerability of multiple doses of two pregabalin controlled release tablets as compared to multiple doses of the pregabalin immediate release capsule.

DETAILED DESCRIPTION:
Evaluate the absorption, pharmacokinetics, safety/tolerability of multiple doses of two pregabalin controlled release tablets as compared to multiple doses of pregabalin immediate release capsule

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve at steady-state over a 24 hour period (AUC24)for assessment of equivalence between 165 mg CR and 75 mg IR (total daily dose 150 mg) | 5 days
AUC24 and maximum plasma concentration over a 24 hour period (Cmax) at steady-state for assessment of equivalence between the 82.5 mg CR (two tablets administered concurrently) and 165 mg CR | 5 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Chew ML, Alvey CW, Plotka A, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pregabalin controlled-release pharmacokinetics in healthy volunteers: analysis of four multiple-dose randomized clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):627-37. doi: 10.1007/s40261-014-0221-2. PMID 25078977
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081226&StudyName=An%20Investigation%20Of%20The%20Absorption%20And%20Pharmacokinetics%20Of%20Multiple%20Doses%20Of%20Two%20Controlled%20Release%20Pregabalin%20Tablets%20As%20Compared%20To%20Mu